CLINICAL TRIAL: NCT03414333
Title: The Effect of Glucagon-like Peptide-1 (GLP-1) on Cognitive and Non-cognitive Function in Human
Brief Title: To Determine the Effect of GLP1 on Cognitive Function, Brain Glucose Metabolism and Neuroplasticity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Stefano Del Prato, Clinical Resercher, University of Pisa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRA 2016
Record Dates: First submitted 2018-01-15; First posted 2018-01-29 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Glucose Metabolism Disorders; Obesity; Degenerative Brain Disorder
Keywords: obesity; cognitive dysfunction
MeSH Terms: conditions — Glucose Metabolism Disorders; Obesity; Cognitive Dysfunction | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roux-en- Y gastric bypass (RYGB) (Experimental): Roux-en- Y gastric bypass (RYGB) is the most popular bariatric procedure and it has been associated with improvements in glycemic control and cognitive function. It works by decreasing the amount of food you can eat at one sitting and by changing the hormones released at the bottom of the stomach and duodenum.we propose that RYGB is a model of chronic elevation of GLP-1 providing an opportunity to explore relationship between changes in the circulating hormone and brain glucose metabolism, cognitive function and neuroplasticity.
  Interventions: Procedure: RYGB
- GLP-1 (Active Comparator): GLP-1 is an intestinal hormone secreted in response to nutrients.
  Interventions: Drug: GLP-1

INTERVENTIONS:
Procedure: RYGB — RYGB is associated with a increase of circulating GLP-1 (up to ten-fold) especially in response to meal ingestion. This increased availability of GLP1 has been claimed to contribute to restoration of some of the beta-cell function.
  Arms: Roux-en- Y gastric bypass (RYGB)
Drug: GLP-1 — GLP-1 is an hormone secreted by gut in response to nutrients ingestion.
  Other Names: gut hormone
  Arms: GLP-1

SUMMARY:
To test the hypothesis that GLP1 can exert favourable effects on multiple aspects of brain function. To this purpose, the investigator determine whether chronic increase in GLP1 concentration as it occurs after bariatric surgery (Roux-en- Y Gastric Bypass) is associated with improvement in:

* cognitive function measured by Mini Mental State Examination (MMSE) and Mental Deterioration Battery(MDB).
* brain glucose metabolism measured by FDG-CT/PET
* neuroplasticity measure by binocular rivalry and saccadic adaptation tests in morbid obese subjects. In order to discern the effect of GLP1 irrespective of changes in the metabolic milieu the investigator will test whether short-term GLP-1 infusion can modulate the same parameters in healthy subjects.

DETAILED DESCRIPTION:
The research project will include two separate studies:

1. In obese subjects undergoing RYGB to test the effect of chronic elevation of GLP1 levels, and
2. In normal volunteers to test the acute effect of GLP1, irrespective of changes in the metabolic milieu In several aspects of brain function as detailed below:.

Morbid Obese Subjects Group:

This study will consist in a single arm, non randomized, uncontrolled, single center before-and after RYGB in 15 morbid obese subjects.

Healthy Subjects Group:

This study will consist in a single arm, non randomized, uncontrolled, single center study in 8 healthy subjects.

The primary endpoint are the changes in:

* cognitive function measured by Mini Mental State Examination (MMSE) and Mental Deterioration Battery (MDB)
* brain glucose metabolism measured by FDG-CT/PET
* neuroplasticity measure by binocular rivalry and saccadic adaptation tests six months after RYGB in morbid obese subjects and with elevation of circulating GLP1 levels in healthy subjects.

Morbid obese subjects participating in this study will be evaluated before and 6 months after bariatric surgery which is routinely performed to treat morbid obesity. For the purpose of baseline assessment subjects will undergo 3 visits at 1 week interval. All test procedures will be repeated in two subsequent visits 6 months after surgery with body weight being stable. Therefore, participation in the study will require a total of 5 visit with a post-trial phone contact 2 weeks after completion for safety assessment.

Healthy subjects will be recruited for determining the acute effect of GLP1 on brain function irrespective of changes in the metabolic milieu. The study will require participation in a total of 3 visits.

ELIGIBILITY:
Inclusion Criteria:(Morbid Obese Subjects Group)

1. Males and females undergoing bariatric surgery as per clinical management
2. Age = 18-60 years
3. BMI>35 Kg/m 2 and stable weight (± 3 lbs) over the preceding three months
4. Normal Glucose Tolerance (HbA1c > 4.5 % and < 5.7%) or Type 2 diabetes (HbA1c >5.7 % and <10.0%)
5. Stable eGFR (>60 ml/min/1.73 m2 )
6. Drug naive for type 2 diabetes treatment or on stable dose more than 3 months with anti-diabetic agents other than DPP4-inhibitors, GLP1 receptor agonists, and insulin.
7. Subjects are capable of giving informed consent

Inclusion Criteria (Healthy Subjects Group)

1. Males and females
2. Age = 18-60 years
3. BMI 22-35 Kg/m 2 and stable weight (± 3 lbs) over the preceding three months
4. Stable eGFR (>60 ml/min/1.73 m 2 )
5. Normal Glucose Tolerance (HbA1c>4.5 % and< 5.7%)
6. Subjects are capable of giving informed consent.

Exclusion Criteria:(both groups)

1. Steroids treatment
2. Psychiatric Disorders
3. Mental Retardation
4. Severe cognitive Impairment
5. Neurodegenerative diseases
6. Epilepsy
7. Depression Treatment
8. Traumatic Brain Injury over the preceding six months
9. Liver function enzymes higher more than two times the upper limit
10. Heart Failure (NYHA III-IV)
11. Type 1 Diabetes
12. Diabetic Ketoacidosis
13. GFR<60 ml/min/1.73 m 2
14. Donation of blood to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 8 weeks prior to the enrollment visit and at least 8 weeks thereafter
15. Women who are pregnant or breastfeeding
16. Patient with a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance which, in the opinion of the investigator or coordinator, might pose an unacceptable risk to the patient or interfere with trial procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
sustained Weight Loss | 6 months
  normalizing obesity-related comorbidities.

SECONDARY OUTCOMES:
glycemic Control | 6 months
  GLP-1 level controled

OTHER OUTCOMES:
cognitive Function | 6 months
  cognitive function measured by Mini Mental State Examination (MMSE).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Del Prato, MD, Principal Investigator — University of Pisa
Locations (1):
- Dept.Clinical and Experimental Medicine.Section of Diabetes., Pisa, Italy

REFERENCES:
- [Derived] Dardano A, Aghakhanyan G, Moretto C, Ciccarone A, Bellini R, Sancho Bornez V, Ceccarini G, Santini F, Volterrani D, Del Prato S, Daniele G. Brain effect of bariatric surgery in people with obesity. Int J Obes (Lond). 2022 Sep;46(9):1671-1677. doi: 10.1038/s41366-022-01162-8. Epub 2022 Jun 21. PMID 35729365